CLINICAL TRIAL: NCT04359056
Title: Integration of Clinical Pharmacy Along the Entire Care Pathway of Patients Implanted with a PICC-line
Brief Title: Clinical Pharmacy for Patients with a PICC Line
Acronym: CLIPICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RC31/18/0459; 2019-A02475-52 (Other: ID RCB)
Record Dates: First submitted 2020-04-08; First posted 2020-04-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Catheter Complications
Keywords: Pharmacists; Equipment and Supplies; Peripheral Catheterization; Operating Rooms; Hospital; Primary Health Care; Medical devices; PICC lines; clinical pharmacy; effectiveness; patient care management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): patients for the observational phase. This corresponds to usual cares where no clinical pharmacy activities will be performed
- Interventional (Experimental): patients for the interventional phase where clinical pharmacy activities will be performed at each step of the care pathway: from hospitalization to home care.
  Interventions: Other: Clinical pharmacy activities along the care pathways

INTERVENTIONS:
Other: Clinical pharmacy activities along the care pathways — PICC line implantation: Optimize the logistics circuit of the PICC line by rationalizing orders through the evaluation of potential losses.
  Ensure the due traceability of the implanted medical device. Discharge order : Analysis, optimization and pharmaceutical interventions if necessary Discharge Pharmaceutical Interview : Discussion with the patient, Information about the PICC line maintenance and associated therapies, Information about the prescribed drugs.
  Call to the community pharmacist to transfer the patient's prescription. Follow-up calls for 3 months after discharge
  * Patients: Two calls the first week after implantation, then one call per month for a maximum of 3 months, Clinical data collection :Pharmaceutical advices if necessary
  * Liberal nurses: same frequency, Clinical data collection, Pharmaceutical advices if necessary
  * Community pharmacist: one call per month, information relevant to the patient's follow-up will be collected.
  Arms: Interventional

SUMMARY:
Clinical pharmacy is a patient-centered discipline and improves significantly the safety of drug management. Regarding medications, clinical pharmacy is efficient. The investigator hypothesize that clinical pharmacy applied to medical devices could be as effective as in the medication field.

The main objective of this study is to assess the effectiveness of clinical pharmacy activities during entire care pathways of patients implanted with a PICC line, in preventing complications.

DETAILED DESCRIPTION:
This is a preliminary, before-after, monocentric and prospective study. The study will begin with an observational period and will be followed by an experimental intervention period. Sixty-nine adult patients in each period will be included. During the observational phase, no clinical pharmacy activities will be performed. During the interventional phase, clinical pharmacists will be active during the entire patients' care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age equal to or older than 18 years old
* Patient capable of giving free and informed consent
* Patient insured by the Social Security System
* Patient living at home
* Patient with a PICC line prescription
* Patient whose discharge prescription should contain drugs and MDs
* Patient for home discharge implanted with a PICC line
* Patient reachable by phone

Exclusion Criteria:

* Under aged patient, age under 18 years old
* Uninsured patient by the Social Security System
* Patient not living at home :
* Institutionalized patient
* Patient living in a home for elderly dependent persons
* Nursing home resident
* Home-hospitalized patient
* Patient deprived of liberty by a judicial or administrative decision
* Patient under guardianship, curatorship or safeguard of justice
* Patient unreachable by phone
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the number of complications during the interventional phase. | 3 months
  Number of complications per patient and per month in each group. Number of complications per patient and per month in each group

SECONDARY OUTCOMES:
Number of consultations and rehospitalizations post-discharge. | 3 months
  Rates of consultations and rehospitalizations in each group.
Acceptance rate of pharmaceutical interventions (PI) during interventional phase and evaluation of PIs' criticality. | 3 months
  Number of potentially inappropriate prescriptions resulting in an accepted PI over total of PIs.
Conformity analysis of the PICC line logistic circuit | day 0
  Number of correct items over total (items checklist about stock, supply chain, traceability)
Conformity analysis of treatment indication. | day 0
  Number of correct items over total (items checklist about recommended indications, implantation duration, etc.)
Conformity analysis of hospital prescriptions issued in town. | day 0
  Conformity rates per phase.
Patient's Quality Of Life assessment | at discharge
  EQ-5D-5L score
Patient's Quality Of Life assessment | 3 months
  EQ-5D-5L score
Participants satisfaction survey | 3 months
  Assessment of patients' satisfactions regarding their therapeutic management
healthcare professionals satisfaction survey | 3 months
  assessment of healthcare professionals' satisfactions regarding their collaboration with the pharmacists
Direct hospital costs. | 3 months
  description and evaluation of the direct medical costs

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte ROUZAUD LABORDE, Principal Investigator — : Institute of metabolic and cardiac diseases (I2MC), Inserm 1048 unit.
Locations (1):
- CIVADE, Toulouse, Occitanie, France

REFERENCES:
- [Derived] Pouget AM, Civade E, Cestac P, Rouzaud-Laborde C. From hospitalisation to primary care: integrative model of clinical pharmacy with patients implanted with a PICC line-research protocol for a prospective before-after study. BMJ Open. 2021 Apr 7;11(4):e039490. doi: 10.1136/bmjopen-2020-039490. PMID 33827827